CLINICAL TRIAL: NCT00056186
Title: Exploration of Transitional Life Events in Individuals With Friedreich's Ataxia: Implications for Genetic Counseling
Brief Title: Transitional Life Events in Patients With Friedreich's Ataxia: Implications for Genetic Counseling
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030118; 03-HG-0118
Record Dates: First submitted 2003-03-07; First posted 2003-03-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-01

CONDITIONS: Friedreich Ataxia
Keywords: Adaptation; Neurodegenerative; Health Care Provider; Psychosocial; Chronic Illness/Disability; Friedreich's Ataxia; Friedreich Ataxia; FA
MeSH Terms: conditions — Friedreich Ataxia; Chronic Disease

SUMMARY:
The purposes of this study are to learn about significant life changes for people with Friedreich's ataxia and about patients' experiences with health care providers. Friedreich's ataxia is a rare genetic disorder in which patients experience progressive muscle weakness and loss of coordination in the arms and legs. They may have other complications, such as vision and hearing impairment, dysarthria, scoliosis, diabetes, and heart disease. The study will explore the impact of this chronic progressive illness on transitional life events, such as career choice and marriage, and the role of family members and health care providers-particularly genetic counselors-in helping patients progress through these events.

Patients with Friedreich's ataxia who are 18 years of age or older may be eligible for this study. Those enrolled will participate in a 45- to 60-minute interview by phone or in person, in which they will be asked questions about important changes in their lives and their past experiences with health care providers. The interview will be audiotaped.

DETAILED DESCRIPTION:
Human development across the lifespan is a process of continual change, adaptation and growth. Throughout this process, key transitional events, such as career choice and marriage, mark important points in time when an individual's life course is significantly altered. These transitional events may be instigated by age, historical or idiosyncratic factors. Of particular interest in the present study are patients' perceptions of transitional events brought about or altered by chronic illness and disability. Additionally, factors (i.e. social support, communication, family) that help facilitate progression through these events will be investigated. The actual or potential role of health care providers during transitional events will also be explored with a specific emphasis on genetic counseling. These themes will be examined through the administration of a one-time, semi-structured, in-person or telephone interview of patients with Friedreich's ataxia: a progressive, debilitating, neurodegenerative condition. The interviews will be approximately 45-60 minutes in length and will include open-ended questions to elicit qualitative data. Approximately 40 subjects will be recruited from Friedreich's ataxia support groups, a research organization and a clinical setting.

It is anticipated that data elicited from the study will lead to recommendations regarding the process and content of genetic counseling for individuals with Friedreich's ataxia. These considerations, coupled with qualitative data obtained from participants, may also have implications for the evolving role of the genetic counselor. Specifically, consideration of developmental counseling approaches, which emphasize key transitional events, may be particularly useful as genetic counselors become increasingly involved in subspecialties (i.e. cardiology, pediatrics, neurology) that provide continuing follow-up care to patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Any individual diagnosed with Friedreich's ataxia, 18 years of age or older, who speaks English and is either in attendance at the NAF conference, or who has access to a telephone.

EXCLUSION CRITERIA:

Adolescents and children under the age of 18. Children and adolescents will be excluded due to the potiential for increased psychological and/or emotional.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-03; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Beisecker AE, Cobb AK, Ziegler DK. Patients' perspectives of the role of care providers in amyotrophic lateral sclerosis. Arch Neurol. 1988 May;45(5):553-6. doi: 10.1001/archneur.1988.00520290089019. PMID 3358709
- [Background] Bernhardt BA, Biesecker BB, Mastromarino CL. Goals, benefits, and outcomes of genetic counseling: client and genetic counselor assessment. Am J Med Genet. 2000 Sep 18;94(3):189-97. doi: 10.1002/1096-8628(20000918)94:33.0.co;2-e. PMID 10995504
- [Background] Borreani C, Gangeri L. Genetic counselling: communication and psychosocial aspects. Tumori. 1996 Mar-Apr;82(2):147-50. doi: 10.1177/030089169608200209. PMID 8644377